CLINICAL TRIAL: NCT04903782
Title: Assessment of the Utility of Family-based (Trio) Whole-genome Sequencing for Cancer Predisposition Testing in Sequential Newly Diagnosed Paediatric and Adolescent Cancer Patients
Brief Title: Cancer Predisposition Testing by Family-based Whole-genome Sequencing (WGS) in Every Child With Newly Diagnosed Cancer
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: Sydney Children's Hospitals Network (Other)
Collaborators: Children's Cancer Institute Australia (Unknown)
Responsible Party: Principal Investigator, Kathy Tucker, Professor, Sydney Children's Hospitals Network
Other Study IDs: PREDICT
Record Dates: First submitted 2021-03-16; First posted 2021-05-27 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Neoplastic Syndromes, Hereditary; Cancer; Genetic Predisposition to Disease
Keywords: Germ-line Mutation; Disease Susceptibility; Child; Pediatrics; Genomics; Next Generation Sequencing; Risk
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Neoplasms; Genetic Predisposition to Disease; Disease Susceptibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with newly diagnosed malignancy
  Interventions: Diagnostic Test: Family-based whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Family-based whole genome sequencing — 1. Germline whole-genome family-based sequencing and variant identification.
  2. Multidisciplinary Meeting case discussion.
  3. Recommendation of referral to a Cancer Genetics Clinic for further investigation, follow up and/or genetic counselling.
  4. Psychosocial study to analyse the impact of germline sequencing on families.

SUMMARY:
Assessment of the utility of family-based (trio) whole-genome sequencing for cancer predisposition testing in sequential newly diagnosed paediatric and adolescent cancer patients

DETAILED DESCRIPTION:
Cancer Predisposition Syndromes (CPS), caused by germline mutations in cancer predisposition genes (CPG) are heritable disorders associated with an increased risk of developing certain types of cancer.

Knowledge of CPG will advance the understanding of tumorigenesis, improve patient care, and facilitate genetic counselling of patients and families. But the prevalence of CPS in Australian children with cancer and the psychosocial impact of germline sequencing to identify CPG have not been studied.

The clinical benefit of family-based WGS in every new child with cancer compared with conventional predictive factors is currently unknown. By testing every child with newly diagnosed cancer the aim is to determine the utility of this approach and its impact on participants and families.

The principal objective of the proposed multicentre prospective study is establish the clinical benefit and utility of family-based WGS to identify underlying CPS in every newly diagnosed child with cancer.

ELIGIBILITY:
* New diagnosis of malignancy
* Age ≤ 21 years
* Written informed consent

Psychosocial component:

* Participants (≥ 12 years)
* Parent/caregiver(s) of participants
* Healthcare professionals involved in the care of patients enrolled in the study

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients who are being treated for a newly diagnosed cancer in New South Wales, Australia
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-03-08 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with CPS identify by WGS as compared to those correctly identified by clinical information (i.e. family history, tumour type, physical findings). | 2 years

SECONDARY OUTCOMES:
The proportion of individuals found to have a reportable germline mutation in a CPG | 2 years
The proportion of patients who have de-novo vs. inherited mutation in CPG. | 2 years
Turnaround time for issuing a report to the treating clinician. | 2 years
The proportion of participants with a complete recording of family history of cancer. | 2 years
Sensitivity and specificity of WGS versus single/multiple gene panel testing guided by clinical predictive factors. | 2 years
The proportion of participants with CPS who undergo cancer surveillance. | 2 years
Test the significance of common cancer risk polymorphisms within a family as a contributing factor in cancer incidence. | 2 years
Quantify the frequency of rare noncoding, complex, and oligogenic variation (in units of variants/person, and genes with variants/person), as detected by WGS, in a paediatric cancer population relative to cancer-free parents and population controls. | 2 years
Assess the prevalence of subclonal somatic variation (e.g. clonal haematopoiesis of indeterminate potential) in children with non-haematological cancer. | 2 years
The psychological impact of the germline sequencing process, including the informed consent process, on patients and parents. | 5 years
  This will be achieved through identifying the incidence of patients and parents enrolled in the study experiencing clinically significant levels of distress, defined as a >7 rating on any of the outcome measures in the Emotion Thermometers Tool©. The incidence of parents and patients experiencing other psychological outcomes such as reduced quality of life will also be identified using the validated scales EuroQoL EQ-5D-5L (parent proxy)/EQ-5D-Y (youth version), Decisional Regret Scale and the Trust In Physician Scale (adapted for a paediatric setting). Psychological outcomes will be re-assessed over the 5 year course of the study to assess impacts of germline sequencing over time.
Cost of clinical model including WGS for cancer predisposition testing in every child newly diagnosed with cancer. | 5 years

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - John Hunter Children's Hospital, Newcastle, New South Wales
  - Sydney Children's Hospital, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuentes Bolanos NA, Padhye B, Daley M, Hunter J, Hetherington K, Warby M, Courtney E, Kirk J, Josephi-Taylor S, Chen Y, Alvaro F, Barlow-Stewart K, Wong-Erasmus M, Barahona P, Ajuyah P, Altekoester AK, Tyrrell VJ, Lau LMS, Wakefield C, Sylvester D, Tucker K, Pinese M, Dalla Pozza L, O'Brien TA. Protocol for a comprehensive prospective cohort study of trio-based whole-genome sequencing for underlying cancer predisposition in paediatric and adolescent patients newly diagnosed with cancer: the PREDICT study. BMJ Open. 2023 May 30;13(5):e070082. doi: 10.1136/bmjopen-2022-070082. PMID 37253493